CLINICAL TRIAL: NCT07346612
Title: Development of the Online Mindfulness-based Intervention (Mind Space Application) for Thai-university Students: Phase II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University (Other)
Responsible Party: Principal Investigator, Chuntana Reangsing, Principal investigator, School of Nursing, Mae Fah Luang University, Thailand, Mae Fah Luang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 25247-19; 692A06004 (Other Grant/Funding Number: Fundamental Fund; FF)
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: University Students; Psychological Well Being; Mindfulness
Keywords: university students; depression; psychological well being
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) collecting all outcomes at baseline and post-intervention by using online web based method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: online mindfulness-based intervention (Experimental): online mindfulness-based intervention The mindfulness-based intervention (mind space) consists of 8 topics, one topic per week. Moreover, the researchers will assign participants (experimental group) to continuously practice using guided meditation approximately 10 minutes daily at least 5 days a week for 3 months via MFU-Mindful application
  Interventions: Behavioral: mind space intervention
- Waitlist control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: mind space intervention — online mindfulness-based intervention The mindfulness-based intervention (MFU-Mindfulapplication) consists of 8 topics, one topic per week.
  Moreover, the researchers will assign participants (experimental group) to continuously practice using guided meditation approximately 10 minutes daily at least 5 days a week for 3 months via MFU-Mindful application
  Arms: Experimental: online mindfulness-based intervention

SUMMARY:
Development of the online mindfulness-based intervention (MFU-mindful Application for Thai university students: Phase II

Objectives:

Phase I: (October 2025 to September 2026)

1. To develop the mindfulness-based intervention (Mind Space application) for Thai university students.
2. To test the feasibility of the mindfulness-based intervention (Mind space Application) for Thai university students.
3. To determine the effect size of mindfulness-based intervention (Mind space Application) on mental health outcomes for Thai university students: A pilot study. Phase II: (October 2026 to December 2026)

1. To examine the effects of mindfulness-base intervention (Mindspace Application) on mental health outcomes for Thai university students For this research project, investigators will develop the mindfulness-based intervention (Mindspace application) based on mindfulness-based stress reduction (MBSR) and mindfulness-based cognitive therapy (MBCT) by encouraging participants to pay attention to their present thoughts, emotions, feelings, and behaviors without judgment. This attention will help them learn the relationship between their thoughts, emotions, and behaviors and their mental health outcomes (mindfulness, stress, anxiety, and depression), though. mindfulness practice (body scan, sitting meditation, and mindful movement) using an online application). Furthermore, investigators will teach participants how to shape their thoughts and manage their wandering minds and negative and irritable thoughts. Finally, participants will learn how to become an individual with reasonable flexibility and positive thoughts.

Settings: the researchers plan to conduct the program in three universities in Northern Thailand.

Population and sample:

Population: Thai university students who are between years 1 and 4 (undergraduate).

Sample:

Phase I: Mae Fah Luang University, Phayao University, and Utraradit University students who are studying during the Fall semester, year 2026. Investigators will specifically recruit volunteers who:

Inclusion criteria:

1. are current studying in years 1-4 of undergraduate programs
2. can read, speak, and write in Thai
3. be risk of the mental health problem (score higher than 6 on the General Health Questionnaire (GHQ-28)
4. have no history of learning disorders (ADHD, other specific learning disorders)
5. have no psychiatric disorders (schizophrenia, adjustment disorders, delusion disorders, and substance use disorders)
6. have no meditation experience within the past 6 months

Exclusion criteria:

1. have a limitation for mindful movement (hearing loss, blindness, and movement limitations)
2. They may feel uncomfortable or distressed and may not be able to participate in each mindfulness-based intervention session.

Conceptual frameworks. For this research project, the investigators will develop and refine an online mindfulness-based intervention, the Mind Space Application, grounded in the principles of Mindfulness-Based Stress Reduction (MBSR; Kabat-Zinn, 2003) and Mindfulness-Based Cognitive Therapy (MBCT; Segal et al., 2002). The program is designed to cultivate nonjudgmental awareness of thoughts, feelings, emotions, and behaviors among university students (Kabat-Zinn, 2003). In addition, it aims to enhance participants' understanding of the interrelationships among cognitions, emotions, affective experiences, and behaviors that contribute to psychological distress, including stress, anxiety, and depressive symptoms.

The intervention incorporates core mindfulness practices delivered via an online application, including body scan exercises, sitting meditation, and mindfulness-based movement for relaxation. Furthermore, participants will be guided to develop cognitive awareness and adaptive responses to internal and external stressors, with particular emphasis on recognizing and managing automatic thoughts (wandering mind), negative thoughts, and irrational or maladaptive cognitions. Through this process, participants are encouraged to cultivate more rational, flexible, and positive thinking patterns.

The researchers anticipate that this program will enhance mindfulness skills and, in turn, contribute to reductions in stress, anxiety, and depressive symptoms among the study participants.

The effectiveness of the Mind Space application will be examined across both short-term and long-term periods. Short-term effects will be assessed at baseline and immediately post-intervention (8 weeks), while long-term effectiveness will be evaluated at a 6-month follow-up. Outcomes in the intervention group will be compared with those in a control group. The primary outcome variables include mental health indicators-stress, anxiety, and depressive symptoms-as well as levels of mindfulness among Thai university students. Data will be analyzed using a one-way repeated-measures multivariate analysis of variance (MANOVA).

ELIGIBILITY:
Inclusion Criteria: the researchers will specifically recruit volunteers who:

1. are current studying in years 1-4 of undergraduate programs
2. can read, speak, and write in Thai
3. be risk of the mental health problem (score higher than 6 on the General Health Questionnaire (GHQ-28))
4. have no history of learning disorders (ADHD, other specific learning disorders)
5. have no psychiatric disorders (schizophrenia, adjustment disorders, delusion disorders, and substance use disorders)
6. have no meditation experience within the past 6 months

Exclusion Criteria: the researchers will exclude the volunteers who;

1. have a limitation for mindful movement (hearing loss, blindness, and movement limitations)
2. uncomfortable or feel distress and cannot participate in each mindfulness-based intervention session

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Suanprung Stress Test-20, SPST-20 | Baseline-at 8 weeks [over 8 week]
  This is a self-administered questionnaire consisting of 20 items, which was adapted and translated into Thai by Mahatnirunkul et al. (1997). This scale provides one score reflecting sensitivity to stress, sources of stress, and physiological reactions to stress (e.g., muscular stress, nervous systems, emotional stress, and cognitive stress). This scale measures how much daily activities produce work-related stress and individuals' responses to stress.
  Respondents are asked to choose from five possible responses in a format requiring them to describe how they feel at this very moment on a 5-point intensity scale: 1 = no stress, 2 = mild stress, 3, = moderate stress, 4 = much stress, and 5=extreme stress. Higher scores indicate higher levels of stress. Researchers have divided the SPST-20 stress scores into four levels: 0-24, mild; 25-42, moderate; 43-62, high; and over 63, severe stress (Mahatnirunkul et al., 1997). Cronbach's alpha was reported to be more than .7
State-Trait Anxiety Inventory Form Y-1 | baseline - 8 week [over 8 wks]
  STAI form -1, Thai version. This scale is a self-report questionnaire developed by Spielberger and Sydeman (1994) and was translated into Thai by Thapinta (1991). This scale consists of 20 items including 10-positive items and 10- negative items. Respondents are asked to choose from four possible responses in a format requiring them to describe how they feel at this very moment on a 4-point intensity scale: 1 = not at all, 2 = somewhat, 3, = moderately, 4 = very much. Thus, possible scores ranged from 1 to 80. Higher scores indicate higher anxiety (Thapinta, 1991). For this study, the Cronbach's alpha coefficient was .80.
Philadelphia Mindfulness Scale, Thai version | baseline- 8 weeks [over 8 weeks]
  This scale is a self-report questionnaire with 20 items, which was developed and translated by Silpakit et al. (2004). It consists of 2 subscales, awareness and acceptance, with response options from 1 to 5 (1=never, 2=rarely, 3=sometimes, 4=often, and 5=very often). A higher score indicates a higher mindfulness level. The Cronbach's alpha coefficient of awareness and acceptance among Thai-population were .87 and .88, respectively (Silpakit et al., 2004). For this study, the Cronbach's alpha coefficient was 0.92 for the total score
Center for Epidemiologic Studies-Depression Scale-Thai version, CES-D-Thai version | baseline - 8 weeks [over 8 wks]
  CES-D Thai version is a self-report questionnaire with a total of 20 items, which was developed by the Center for Epidemiologic Studies at the U.S. National Institute of Mental Health and was translated and adapted into Thai by Trangkasombat et al. (1997). The reliability of this instrument was .86 among Thai adolescents (Trangkasombat et al., 1997). Respondents are asked to choose from four possible responses where 0 = rarely or none of the time (less than 1 day), and 4 = almost or all of the time (5 to 7 days). A total score is calculated by summing all items providing a possible range from 0 to 60. Higher scores reflect greater levels of depressive symptoms. The CES-D has 4 separate subscales: positive affect, negative affect, somatic symptoms, and interpersonal relations. Items on the positive affect subscale are reversed to reflect 'unhappy' or 'lack of well-being' (Trangkasombat et al., 1997). The CES-D has good internal consistency with alphas of 0.85 for the general population

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Mae Fah Luang University, Chiang Rai, Chiangrai, Thailand

IPD SHARING:
Plan to Share IPD: No
Prohibit from law